CLINICAL TRIAL: NCT00150865
Title: Study of Posterior Lumbar Plexus Block for Pain Relief After Hip Surgery
Brief Title: Evaluation of Efficacy of Lumbar Plexus Bloc After Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CP 02-01
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2005-09

CONDITIONS: Pain; Postoperative
Keywords: ropivacaine; posterior lumbar plexus block; hip arthroplasy; analgesia; postoperative
MeSH Terms: conditions — Pain; Agnosia | interventions — Ropivacaine

INTERVENTIONS:
Drug: ropivacaine

SUMMARY:
Compare lumbar plexus block with ropivacaine 0.475%, 0.4 ml/kg to saline. Each group randomized, includes 30 patients. block performed preoperatively Surgery under general anesthesia. Postoperative evaluation of pain (VAS) as first endpoint, and also morphine consumption via PCA device. Follow-up : 24h.

Expectation : sizeable reduction of pain with block, of duration.

DETAILED DESCRIPTION:
Compare lumbar plexus block (randomized)

* ropivacaine 0.475%, 0.4 ml/kg
* saline 0.4 ml/kg . Each group includes 30 patients.

Block performed preoperatively.

Surgery under general anesthesia (sufentanil, propofol, atracurium ; maintenance : sevoflurane and nitrous oxide in O2. Sufentanil added peroperatively as clinically needed.

Postoperative evaluation of pain (VAS, by an independant blind observer) as first endpoint, and also morphine consumption via PCA device.

Adverse effects (nausea, vomiting, etc) recorded

Follow-up : 24h. Expectation : sizeable reduction of pain with block, of duration.

ELIGIBILITY:
Inclusion Criteria:

* adults
* ASA 1-3

Exclusion Criteria:

* cognitive impairement
* ASA IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2001-09; Study Completion 2002-03

PRIMARY OUTCOMES:
decrease of postoperative pain

SECONDARY OUTCOMES:
decrease in morphine consumption
duraration of analgesic effect

CONTACTS AND LOCATIONS:
Overall Officials: laurent beydon, MD, Study Director — University Hospital, Angers; ibrahim okais, MD, Principal Investigator — Clinique St Leonard